CLINICAL TRIAL: NCT02598388
Title: A Randomized, Observer-blind, Placebo-controlled, Two-part, Phase 2 Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Prime-boost Regimens of the Candidate Prophylactic Vaccines for Ebola Ad26.ZEBOV and MVA-BN-Filo
Brief Title: Safety, Tolerability and Immunogenicity Study of 2-dose Heterologous Regimens for Ebola Vaccines Ad26.ZEBOV/MVA-BN-Filo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR108062; VAC52150EBL2003 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Healthy; Vaccine; Ebola viruses; Ebola virus disease (EVD); Filoviruses; Hemorrhagic fever; Monovalent vaccine; Human adenovirus serotype 26 (Ad26) encoding the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic (MVA-BN) Filo-vector; Safety; Immunogenicity
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (US Participants) (Experimental): Participants will receive MVA-BN-Filo or placebo on Day 1 followed by Ad26.ZEBOV or placebo on Day 15.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo
- Part 2 Group 1 (African Participants) (Experimental): Participants will receive Ad26.ZEBOV or placebo on Day 1 followed by MVA-BN-Filo or placebo on Day 29.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo
- Part 2 Group 2 (African Participants) (Experimental): Participants will receive MVA-BN-Filo or placebo on Day 1 followed by Ad26.ZEBOV or placebo on Day 15.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV — One 0.5 mL intramuscular (IM) injection of (5x10*10 viral particles).
Biological: MVA-BN-Filo — One 0.5 mL IM injection of (1x10*8 infectious units).
Biological: Placebo — One 0.5 mL IM injection of 0.9 percent (%) saline.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of different vaccination schedules of Ad26.ZEBOV and MVA-BN-Filo administered intramuscularly (IM) as 2-dose heterologous regimens in healthy and in HIV-infected adults.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, placebo-controlled, parallel-group, multicenter, 2-part, Phase 2 study of Ad26.ZEBOV and MVA-BN-Filo in healthy and HIV infected adults. In part 1, dose 1 vaccination with MVA-Bn-Filo will be followed by dose 2 vaccination with Ad26 14 days later in the US. In part 2, two regimens will be investigated. The first regimen will be Ad26 dose 1 vaccination followed by MVA-BN-Filo dose 2, 28 days later and the second regimen will be MVA-BN-Filo dose 1 vaccination followed by Ad26.ZEBOV dose 2, 14 days later in Africa. The study consists of a Screening phase of up to 8 weeks (starting from the moment the participants signs the ICF), a Vaccination Phase, in which participants will be vaccinated at baseline (Day 1) followed by a dose 2 vaccination on Day 15 or 29, and a post-dose 2 follow-up phase of maximum 1 year post-dose 2 vaccination. Upon completion of 6-month post dose 2 visit those participants who received active vaccine will enter long-term follow-up until the 1 year post dose 2 vaccination visit to assess long-term safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy in the Investigator's clinical judgment on the basis of medical history, physical examination and vital signs performed at Screening
* Participant must be healthy on the basis of clinical laboratory tests and electrocardiogram (ECG) (only in participants >50 years) performed at Screening. If the results of the laboratory screening tests and ECG are outside the institutional normal reference ranges, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study
* A woman of childbearing potential must have a negative urine β-human chorionic gonadotropin [beta-hCG] pregnancy test at Screening and a negative urine [beta-hCG] pregnancy test immediately prior to each study vaccine administration
* A man who is sexually active with a woman of childbearing potential must be willing to use condoms for sexual intercourse beginning prior to dose 1 vaccination until at least 3 months after the dose 2 vaccination, unless a vasectomy was performed more than 1 year prior to Screening
* Participant must pass the test of understanding (TOU)
* Additional Inclusion Criteria for HIV-infected participants a) participants must have a positive HIV-1 and/or -2 serology test within 6 months of screening, including the day of screening; b) participants must have a Screening CD4+ cell count >200 cells/microliter (mcL); c) in part 1, all participants must be on a stable highly active antiretroviral therapy (HAART) regimen for 4 weeks prior to Screening, in part 2 participants with screening CD4+ cell count <350 cells/mcL must also be on a stable HAART regimen for 4 weeks prior to Screening

Exclusion Criteria:

* Has received any candidate Ebola vaccine
* Diagnosed with Ebola virus disease, or prior exposure to EBOV, including travel to epidemic Ebola areas less than 1 month prior to Screening
* Has received any experimental candidate Ad26- or MVA-based vaccine in the past or received any other investigational drug or investigational vaccine or used an invasive investigational medical device within 3 months prior to Screening
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products
* Presence of significant conditions (eg, history of seizure disorders, (auto)immune disease or deficiency, any spleen disease, active malignancy, ongoing tuberculosis treatment, other systemic infections) or clinically significant findings during screening of medical history, ECG (only in participants >50 years), physical examination, vital signs or laboratory testing for which, in the opinion of the investigator, participation would not be in the best interest of the participants (eg, compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (7):
- Silver Spring, Maryland, United States
- Kenya (2):
  - Kericho
  - Kisumu
- Maputo, Mozambique
- Abuja, Nigeria
- Mbeya, Tanzania
- Kampala, Uganda

REFERENCES:
- [Derived] Ake JA, Paolino K, Hutter JN, Cicatelli SB, Eller LA, Eller MA, Costanzo MC, Paquin-Proulx D, Robb ML, Tran CL, Anova L, Jagodzinski LL, Ward LA, Kilgore N, Rusnak J, Bounds C, Badorrek CS, Hooper JW, Kwilas SA, Ilsbroux I, Anumendem DN, Gaddah A, Shukarev G, Bockstal V, Luhn K, Douoguih M, Robinson C. Safety and Immunogenicity of an Accelerated Ebola Vaccination Schedule in People with and without Human Immunodeficiency Virus: A Randomized Clinical Trial. Vaccines (Basel). 2024 May 4;12(5):497. doi: 10.3390/vaccines12050497. PMID 38793748
- [Derived] Mwesigwa B, Sawe F, Oyieko J, Mwakisisile J, Viegas E, Akintunde GA, Kosgei J, Kokogho A, Ntinginya N, Jani I, Shukarev G, Hooper JW, Kwilas SA, Ward LA, Rusnak J, Bounds C, Overman R, Badorrek CS, Eller LA, Eller MA, Polyak CS, Moodley A, Tran CL, Costanzo MC, Leggat DJ, Paquin-Proulx D, Naluyima P, Anumendem DN, Gaddah A, Luhn K, Hendriks J, McLean C, Douoguih M, Kibuuka H, Robb ML, Robinson C, Ake JA. Safety and Immunogenicity of Accelerated Heterologous 2-Dose Ebola Vaccine Regimens in Adults With and Without HIV in Africa. Clin Infect Dis. 2024 Oct 15;79(4):888-900. doi: 10.1093/cid/ciae215. PMID 38657084

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 578 randomized participants, 574 received at least one dose of study vaccine.
Groups:
- Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants): Healthy participants received an intramuscular (IM) injection of a single dose MVA-BN-Filo (Dose 1) at Day 1 followed by an IM injection of a single dose Ad26.ZEBOV (Dose 2) at Day 15.
- Part 1: Placebo (Healthy Participants); Part 2 (Group 2): Placebo (Healthy Participants): Healthy participants received an IM injection of a single dose placebo (Dose 1) at Day 1 followed by an IM injection of a single dose placebo (Dose 2) at Day 15.
- Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants): Human immunodeficiency virus (HIV) infected participants received an IM injection of a single dose MVA-BN-Filo (Dose 1) at Day 1 followed by an IM injection of a single dose Ad26.ZEBOV (Dose 2) at Day 15.
- Part 1: Placebo (HIV-infected Participants); Part 2 (Group 2): Placebo (HIV-infected Participants): HIV-infected participants received an IM injection of a single dose placebo (Dose 1) at Day 1 followed by an IM injection of a single dose placebo (Dose 2) at Day 15.
- Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants): Healthy participants received an IM injection of a single dose Ad26.ZEBOV (Dose 1) at Day 1 followed by an IM injection of a single dose MVA-BN-Filo (Dose 2) at Day 29.
- Part 2 (Group 1): Placebo (Healthy Participants): Healthy participants received an IM injection of a single dose placebo (Dose 1) at Day 1 followed by an IM injection of a single dose placebo (Dose 2) at Day 29.
- Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants): HIV-infected participants received an IM injection of a single dose Ad26.ZEBOV (Dose 1) at Day 1 followed by an IM injection of a single dose MVA-BN-Filo (Dose 2) at Day 29.
- Part 2 (Group 1): Placebo (HIV-infected Participants): HIV-infected participants received an IM injection of a single dose placebo (Dose 1) at Day 1 followed by an IM injection of a single dose placebo (Dose 2) at Day 29.
- Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants): Healthy participants received an IM injection of a single dose MVA-BN-Filo (Dose 1) at Day 1 followed by an IM injection of a single dose Ad26.ZEBOV (Dose 2) at Day 15.
- Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants): HIV-infected participants received an IM injection of a single dose MVA-BN-Filo (Dose 1) at Day 1 followed by an IM injection of a single dose Ad26.ZEBOV (Dose 2) at Day 15.
Period: Overall Study
Arm/Group | Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 1: Placebo (Healthy Participants) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 1: Placebo (HIV-infected Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 2 (Group 2): Placebo (Healthy Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 2 (Group 2): Placebo (HIV-infected Participants)
Started | 40 | 10 | 20 | 5 | 161 | 39 | 161 | 39 | 39 | 10 | 40 | 10
Completed | 39 | 10 | 18 | 5 | 151 | 38 | 156 | 38 | 39 | 9 | 39 | 10
Not Completed | 1 | 0 | 2 | 0 | 10 | 1 | 5 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 5 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 1: Placebo (Healthy Participants) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 1: Placebo (HIV-infected Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 2 (Group 2): Placebo (Healthy Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 2 (Group 2): Placebo (HIV-infected Participants) | Total
Number analyzed (Participants) | 40 | 10 | 20 | 5 | 161 | 39 | 161 | 39 | 39 | 10 | 40 | 10 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14.42) | 47.3 (11.84) | 46.7 (12.89) | 46 (8.63) | 29.1 (7.56) | 28.4 (7.37) | 37.5 (9.78) | 38.9 (8.74) | 28 (7.72) | 26.9 (12.56) | 38.5 (9.91) | 41 (9.78) | 34.8 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 2 | 1 | 69 | 19 | 95 | 22 | 20 | 6 | 26 | 4 | 289
  Male | 22 | 3 | 18 | 4 | 92 | 20 | 66 | 17 | 19 | 4 | 14 | 6 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 0 | 7 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 20
  Not Hispanic or Latino | 37 | 10 | 18 | 5 | 154 | 38 | 158 | 37 | 38 | 9 | 40 | 10 | 554
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 6 | 13 | 4 | 160 | 39 | 159 | 39 | 39 | 10 | 40 | 10 | 538
  White | 21 | 4 | 5 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  KENYA | 0 | 0 | 0 | 0 | 50 | 9 | 79 | 21 | 10 | 6 | 15 | 7 | 197
  MOZAMBIQUE | 0 | 0 | 0 | 0 | 32 | 7 | 23 | 5 | 8 | 3 | 5 | 0 | 83
  NIGERIA | 0 | 0 | 0 | 0 | 17 | 3 | 11 | 1 | 2 | 0 | 3 | 1 | 38
  TANZANIA, UNITED REPUBLIC OF | 0 | 0 | 0 | 0 | 31 | 9 | 14 | 4 | 11 | 1 | 4 | 1 | 75
  UGANDA | 0 | 0 | 0 | 0 | 31 | 11 | 34 | 8 | 8 | 0 | 13 | 1 | 106
  UNITED STATES | 40 | 10 | 20 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 75

OUTCOME MEASURES:

1. Primary Outcome: Part 1, Part 2 (Group 2): Number of Participants With Unsolicited Adverse Events
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited adverse events were events which were reported by the participant voluntarily or obtained by means of interviewing the participant in a nondirected manner at study visits. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: Up to 28 days post each dose (up to Day 43)
Population: Safety set was based on full analysis set (FAS) which included all participants who were randomized and received at least 1 dose of study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Groups:
- Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV: Healthy participants in Part 1 and Part 2 (Group 2) received intramuscular (IM) injection of single dose MVA-BN-Filo (Dose 1) on Day 1 followed by IM injection of single dose Ad26.ZEBOV (Dose 2) at Day 15.
- Healthy (Part 1, Part 2; Group 2): Placebo: Healthy participants in Part 1 and Part 2 (Group 2) received IM injection of single dose placebo (Dose 1) on Day 1 followed by IM injection of single dose placebo (Dose 2) at Day 15.
- HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV: Human immunodeficiency virus (HIV)- infected participants in Part 1 and Part 2 (Group 2) received IM injection of single dose MVA-BN-Filo (Dose 1) on Day 1 followed by IM injection of single dose Ad26.ZEBOV (Dose 2) at Day 15.
- HIV-infected (Part 1, Part 2; Group 2): Placebo: HIV-infected participants in Part 1 and Part 2 (Group 2) received IM injection of single dose placebo (Dose 1) on Day 1 followed by IM injection of single dose placebo (Dose 2) at Day 15.
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 79 | 20 | 60 | 15
Participants | 33 | 10 | 32 | 3

2. Primary Outcome: Part 2 (Group 1): Number of Participants With Unsolicited Adverse Events
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited adverse events were events which were reported by the participant voluntarily or obtained by means of interviewing the participant in a nondirected manner at study visits.
Time Frame: Up to 28 days post dose 2 visit (up to Day 57)
Population: Safety set was based on FAS which included all participants who were randomized and received at least 1 dose of study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 161 | 39 | 161 | 39
Participants | 83 | 21 | 78 | 15

3. Primary Outcome: Part 1, Part 2 (Group 2): Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: Up to 1 year post dose 2 (up to Day 380)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV: HIV-infected participants in Part 1 and Part 2 (Group 2) received IM injection of single dose MVA-BN-Filo (Dose 1) on Day 1 followed by IM injection of single dose Ad26.ZEBOV (Dose 2) at Day 15.
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 79 | 20 | 60 | 15
Participants | 1 | 1 | 3 | 1

4. Primary Outcome: Part 2 (Group 1): Number of Participants With SAEs
Description: A SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 1 year post dose 2 (up to Day 394)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 161 | 39 | 161 | 39
Participants | 1 | 1 | 2 | 0

5. Primary Outcome: Part 1, Part 2 (Group 2): Number of Participants With Immediate Reportable Events (IREs)
Description: The following neuroinflammatory disorders were considered immediate reportable events and which had to be reported to the sponsor within 24 hours of becoming aware of the event: cranial nerve disorders including paralyses/paresis (example: bell's palsy), optic neuritis, multiple sclerosis, transverse myelitis, guillain-barre syndrome including miller fisher syndrome, bickerstaff's encephalitis and other variants, acute disseminated encephalomyelitis, including site-specific variants (example: non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis), myasthenia gravis and lambert-eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, including chronic inflammatory, demyelinating polyneuropathy, multifocal motor neuropathy, and polyneuropathies associated with monoclonal gammopathy, narcolepsy, isolated paresthesia of more than 7 days duration.
Time Frame: Up to 1 year post dose 2 (up to Day 380)
Population: Safety set was based on FAS which included all participants who were randomized and received at least 1 dose of study vaccine, regardless of the occurrence of protocol deviations. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 79 | 20 | 60 | 15
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Part 2 (Group 1): Number of Participants With IREs
Description: as for outcome 5
Time Frame: Up to 1 year post dose 2 (up to Day 394)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 161 | 39 | 161 | 39
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Parts 1 and 2: Number of Participants With Solicited Local Adverse Events (AEs) 7 Days Post First Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post first vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: 7 days post dose 1 (up to Day 8)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 79 | 20 | 60 | 15 | 161 | 39 | 161 | 39
Participants | 46 | 5 | 34 | 3 | 71 | 10 | 75 | 7

8. Primary Outcome: Part 1, Part 2 (Group 2): Number of Participants With Solicited Local AEs 7 Days Post Second Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post second vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: 7 days post dose 2 (up to Day 22)
Population: Safety set was based on FAS which included all participants who were randomized and received at least 1 dose of study vaccine, regardless of the occurrence of protocol deviations. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 78 | 20 | 58 | 14
Participants | 44 | 4 | 33 | 0

9. Primary Outcome: Part 2 (Group 1): Number of Participants With Solicited Local AEs 7 Days Post Second Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post second vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site.
Time Frame: 7 days post dose 2 (up to Day 36)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 159 | 37 | 160 | 38
Participants | 82 | 7 | 64 | 7

10. Primary Outcome: Parts 1 and 2: Number of Participants With Solicited Systemic Adverse Events 7 Days Post First Vaccination
Description: Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: 7 days post dose 1 (up to Day 8)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 79 | 20 | 60 | 15 | 161 | 39 | 161 | 39
Participants | 39 | 10 | 37 | 7 | 109 | 24 | 97 | 18

11. Primary Outcome: Part 1, Part 2 (Group 2): Number of Participants With Solicited Systemic AEs 7 Days Post Second Vaccination
Description: as for outcome 10
Time Frame: 7 days post dose 2 (up to Day 22)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 78 | 20 | 58 | 14
Participants | 45 | 8 | 35 | 4

12. Primary Outcome: Part 2 (Group 1): Number of Participants With Solicited Systemic AEs 7 Days Post Second Vaccination
Description: Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Time Frame: 7 days post dose 2 (up to Day 36)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 159 | 37 | 160 | 38
Participants | 83 | 20 | 80 | 10

13. Primary Outcome: Part 1, Part 2 (Group 2): Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against Ebola Virus Glycoprotein (EBOV GP) Measured Using Filovirus Animal Non-Clinical Group (FANG) Enzyme-linked Immunosorbent Assay (ELISA)
Description: GMCs of antibodies binding to EBOV GP using FANG ELISA were reported and were measured in ELISA unit per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using FANG ELISA to determine humoral responses following vaccination. A sample was considered positive, if the value was above the lower limit of quantification (LLOQ), that is, 36.11 ELISA units/mL. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts.
Time Frame: 21-days post dose 2 (up to Day 36)
Population: The per protocol analysis set included all randomized and vaccinated participants, who received both the dose 1 and dose 2 vaccinations (administered within the protocol-defined visit window), had at least 1 post-vaccination (that is, after the date of vaccination) evaluable immunogenicity sample, and had no major protocol violations influencing the immune responses. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Healthy (Part 1, Part 2; Group 2): Placebo | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): Placebo
Number analyzed (Participants) | 68 | 18 | 56 | 13
EU/mL | 5733 [4245 to 7742] | 40 [NA to 112] — Here, 'NA' signifies that lower limit of calculated 95% CI was less than LLOQ. | 2325 [1632 to 3313] | NA [NA to 38] — Here, 'NA' signifies that geometric mean and lower limit of calculated 95% CI was less than LLOQ.

14. Primary Outcome: Part 2 (Group 1): GMCs of Binding Antibody Levels Against EBOV GP Measured Using FANG ELISA
Description: GMCs of antibodies binding to EBOV GP using FANG ELISA were reported and were measured in ELISA unit per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using FANG ELISA to determine humoral responses following vaccination. A sample was considered positive, if the value was above the LLOQ, that is, 36.11 ELISA units/mL.
Time Frame: 21-days post dose 2 (Day 50)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
Number analyzed (Participants) | 151 | 34 | 155 | 36
EU/mL | 6037 [4996 to 7297] | NA [NA to NA] — Here, "NA" signifies that calculated Geometric mean and the limits of the 95% CI were less than LLOQ | 2939 [2316 to 3729] | NA [NA to NA] — Here, "NA" signifies that calculated Geometric mean and the limits of the 95% CI were less than LLOQ

15. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. As per planned analysis, the data from Parts 1 and 2 (Group 2) of the study was pooled (that is, 14-day interval regimen) and presented separately for the healthy and HIV-infected cohorts. This outcome measure was planned to compare the safety (unsolicited AEs, solicited local and solicited systemic AEs) of Ad26.ZEBOV/MVA-BN-Filo and MVA-BN-Filo/Ad26.ZEBOV regimens in healthy and HIV-infected participants. Therefore, placebo arm is not reported.
Time Frame: Solicited AEs: Up to 7 days post each vaccination (Up to Day 36); Unsolicited AEs: Up to 28 days post each vaccination (Up to Day 57)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV: Healthy participants in Part 1 and Part 2 (Group 2) received intramuscular (IM) injection of single dose MVA-BN-Filo as prime vaccine on Day 1 followed by IM injection of single dose Ad26.ZEBOV as booster vaccine at Day 15.
- HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV: HIV-infected participants in Part 1 and Part 2 (Group 2) received IM injection of single dose MVA-BN-Filo as prime vaccine on Day 1 followed by IM injection of single dose Ad26.ZEBOV as booster vaccine at Day 15.
Arm/Group | Healthy (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | HIV-infected (Part 1, Part 2; Group 2): MVA-BN-Filo and Ad26.ZEBOV | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants)
Number analyzed (Participants) | 79 | 60 | 161 | 161
Participants
  Unsolicited AEs | 33 | 32 | 83 | 78
  Solicited Local AEs | 56 | 47 | 103 | 93
  Solicited Systemic AEs | 56 | 46 | 116 | 117

ADVERSE EVENTS:
Time Frame: Up to Day 380 (Part 1, Part 2; Group 2) and Up to Day 394 (Part 2; Group 1)
Description: Safety set included all participants who were randomized and received at least 1 dose of study vaccine, regardless of the occurrence of protocol deviations.
Arm/Group | Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 1: Placebo (Healthy Participants) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 1: Placebo (HIV-infected Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) | Part 2 (Group 2): Placebo (Healthy Participants) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) | Part 2 (Group 2): Placebo (HIV-infected Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) | Part 2 (Group 1): Placebo (Healthy Participants) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) | Part 2 (Group 1): Placebo (HIV-infected Participants)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/10 | 0/20 | 0/5 | 0/39 | 0/10 | 0/40 | 0/10 | 0/161 | 0/39 | 0/161 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/10 | 1/20 | 1/5 | 0/39 | 0/10 | 2/40 | 0/10 | 1/161 | 1/39 | 2/161 | 0/39
Other Adverse Events (participants affected / at risk) | 11/40 | 5/10 | 11/20 | 0/5 | 12/39 | 5/10 | 13/40 | 3/10 | 53/161 | 15/39 | 51/161 | 11/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) (N=40) | Part 1: Placebo (Healthy Participants) (N=10) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) (N=20) | Part 1: Placebo (HIV-infected Participants) (N=5) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) (N=39) | Part 2 (Group 2): Placebo (Healthy Participants) (N=10) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) (N=40) | Part 2 (Group 2): Placebo (HIV-infected Participants) (N=10) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) (N=161) | Part 2 (Group 1): Placebo (Healthy Participants) (N=39) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) (N=161) | Part 2 (Group 1): Placebo (HIV-infected Participants) (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) (N=40) | Part 1: Placebo (Healthy Participants) (N=10) | Part 1: MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) (N=20) | Part 1: Placebo (HIV-infected Participants) (N=5) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (Healthy Participants) (N=39) | Part 2 (Group 2): Placebo (Healthy Participants) (N=10) | Part 2 (Group 2): MVA-BN-Filo and Ad26.ZEBOV (HIV-infected Participants) (N=40) | Part 2 (Group 2): Placebo (HIV-infected Participants) (N=10) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (Healthy Participants) (N=161) | Part 2 (Group 1): Placebo (Healthy Participants) (N=39) | Part 2 (Group 1): Ad26.ZEBOV and MVA-BN-Filo (HIV-infected Participants) (N=161) | Part 2 (Group 1): Placebo (HIV-infected Participants) (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Injection Site Erosion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0 | 5 | 1 | 5 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 5 | 3 | 3 | 3 | 23 | 4 | 25 | 5
Apheresis Related Complication (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 3 | 4 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 9 | 3 | 9 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT02598388/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT02598388/SAP_001.pdf